CLINICAL TRIAL: NCT00025857
Title: Adolescent Medial Temporal Lobe Function in Health and Illness
Brief Title: Brain Function in Mentally Ill Adolescents
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020007; 02-M-0007
Record Dates: First submitted 2001-10-26; First posted 2001-10-29 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2012-06-29

CONDITIONS: Healthy; Posttraumatic Stress Disorder; Major Depressive Disorder
Keywords: fMRI; Depression; PTSD; Emotion; Magnetic Resonance Imaging; Anxiety; Normal Volunteers; Adolescence; Memory; Physical/Sexual Abuse History; Post-Traumatic Stress Disorder; Adolescent; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Depression; Anxiety Disorders

SUMMARY:
The purpose of this study is to use brain imaging technology to examine the brain activity of adolescents with post-traumatic stress disorder (PTSD) and/or major depressive disorder (MDD) before and after treatment.

Adults with PTSD or MDD exhibit abnormalities in the structure and function of certain parts of the brain. Although PTSD and MDD are psychiatric disorders that often emerge in childhood, the relationship between these disorders and brain structures has not been thoroughly studied in adolescents with the disorders. This study will use functional magnetic resonance imaging (fMRI) to study the parts of the brain that are involved in PTSD and MDD in adolescents.

Adolescents with PTSD and/or MDD will be enrolled along with healthy adolescents with or without a history of abuse. Healthy adults will also be enrolled. Participants will be screened with a physical examination; blood tests; and interviews about mood, general degree of nervousness, and behavior. Adolescents and their parents will be interviewed separately and together. Following the interviews, participants will undergo psychological tests. Participants with PTSD and/or MDD will have two weekly sessions of talk therapy. Participants who continue to experience PTSD or MDD symptoms after the talk therapy may continue the talk therapy alone, begin treatment with fluoxetine (Prozac ) alone, or begin fluoxetine in addition to the talk therapy. Participants who take fluoxetine will have blood collected before treatment and 8 weeks after treatment has begun. If participants do not respond to the treatment, the treatment will be stopped and the participants will be offered another treatment. Participants who respond to treatment will continue treatment at NIH until a referral to an outside physician is made. Depending on the experiment in which they are enrolled, participants will undergo one or four MRI scans. Participants who will have four MRI scans will undergo the scans on separate days. During the MRI, participants will complete tasks on a computer. Saliva samples will be collected before and after the scans. Participants with PTSD and/or MDD will collect their saliva one or two days before the MRI scan.

DETAILED DESCRIPTION:
Adults with post-traumatic stress disorder (PTSD) or major depressive disorder (MDD) exhibit abnormalities in the structure and function of the amygdala and hippocampus (temporal lobe), as well as in the prefrontal cortex (PFC) and striatum (four brain structures underlying the emotional processing and reward systems). However, while these psychiatric disorders often emerge in childhood, the integrity of these neural structures has been minimally studied in psychiatrically impaired children and adolescents. In the current proposal, functional MRI (fMRI) will be used to evaluate the amygdala, hippocampus, PFC and striatum in (1) psychiatrically healthy adolescents; (2) adolescents with trauma history and PTSD or anxiety symptoms; (3) adolescents with trauma history, symptoms of depression and either PTSD or anxiety symptoms; and (4) adolescents with only major depressive or PTSD/anxiety symptoms; (5) adolescents with trauma and no trauma related symptoms. The proposed study is conducted in three separate experiments.

At this stage of the protocol, we completed experiment 1, and a pilot study to help guide experiments 2 and 3. In Experiment 1, we determined whether a fear conditioning paradigm elicited amygdala activity in healthy adolescents. The pilot study examined test-retest reliability of the fMRI signal in healthy adolescents and adults.

In Experiment 2, we will examine the functioning of the amygdala, hippocampus, PFC and striatum in healthy adolescents and those with the psychiatric conditions described above. During image acquisition, four cognitive tasks, targeting these regions, will be used: 1) a social interaction task, 2) an inhibition task (the Stop task or the antisaccade task), 3) an emotional rating/explicit memory task and 4) a probe detection task. One hundred twenty five participants (25 in five groups) will be recruited in experiment 2.

Experiment 3 will address the same question as in experiment 2 in relation to treatment response. In other words, in contrast to experiment 2, patients will be studied prior and after treatment of the psychopathology associated with their traumatic experience. The sample will include 125 patients (25 in each of the 4 groups) and 25 controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects 7-18 (adolescents).

Consent: can give consent/assent.

IQ: all subjects will have IQ greater than 70.

Subjects currently on antidepressants or benzodiazepines medication.

Subjects suffering from ADHD and currently on stimulants.

SUBJECTS WITH MAJOR DEPRESSION:

Diagnosis: Current diagnosis of MDD.

Clinical Impairment: CGAS less than 60.

SUBJECTS WITH PTSD:

Diagnosis: current diagnosis of PTSD.

Clinical Impairment: CGAS of less than 60.

SUBJECTS WITH HISTORY OF TRAUMA:

Trauma (i.e., sexual or physical abuse, exposure to an accident, etc.) will be defined according to the KSADS, the Child Trauma Questionnaire, the Life Events Survey and the history of adoption.

EXCLUSION CRITERIA:

Any medical condition that increases risk for MRI (e.g. pacemaker, metallic foreign material in eye).

Any medical condition that increases risk for fluoxetine treatment for patients with MDD/PTSD.

Pregnancy.

Participants suffering from acute psychosis or suicidal ideation; current abuse/dependency to alcohol or drugs.

Currently in an abusive situation at home.

Weight that is 15% more or less than ideal body weight for sex and height.

Current tobacco use.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2001-10-22; Study Completion 2012-06-29

CONTACTS AND LOCATIONS:
Overall Officials: Monique Ernst, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernstein DP, Fink L, Handelsman L, Foote J, Lovejoy M, Wenzel K, Sapareto E, Ruggiero J. Initial reliability and validity of a new retrospective measure of child abuse and neglect. Am J Psychiatry. 1994 Aug;151(8):1132-6. doi: 10.1176/ajp.151.8.1132. PMID 8037246
- [Background] Birmaher B, Dahl RE, Ryan ND, Rabinovich H, Ambrosini P, al-Shabbout M, Novacenko H, Nelson B, Puig-Antich J. The dexamethasone suppression test in adolescent outpatients with major depressive disorder. Am J Psychiatry. 1992 Aug;149(8):1040-5. doi: 10.1176/ajp.149.8.1040. PMID 1636803
- [Background] Blair RJ, Morris JS, Frith CD, Perrett DI, Dolan RJ. Dissociable neural responses to facial expressions of sadness and anger. Brain. 1999 May;122 ( Pt 5):883-93. doi: 10.1093/brain/122.5.883. PMID 10355673